CLINICAL TRIAL: NCT00563784
Title: A Phase II Study of TARCEVA (Erlotinib) in Combination With Chemoradiation in Patients With Stage IIIA/B Non-Small Cell Lung Cancer (NSCLC)
Brief Title: TARCEVA (Erlotinib) in Combination With Chemoradiation in Patients With Stage IIIA/B Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-1023; NCI-2012-01761 (Registry Identifier: NCI CTRP); W81XWH-05-2-0027 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Non-Small Cell Lung Cancer; Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; Squamous Cell Carcinoma; Adenocarcinoma; Bronchoalveolar Cell Carcinoma; Large Cell Anaplastic Carcinoma; Giant Cell Carcinoma; Clear Cell Carcinoma; Erlotinib; Erlotinib Hydrocholoride; OSI-774; Tarceva; Carboplatin; Paraplatin; Paclitaxel; Taxol; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma, Squamous Cell; Adenocarcinoma; Carcinoma, Giant Cell; Adenocarcinoma, Clear Cell | interventions — Erlotinib Hydrochloride; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erlotinib + Paclitaxel + Carboplatin (Experimental): Oral Erlotinib 150 mg daily + Paclitaxel 45 mg/m^2 by vein weekly + Carboplatin 2 AUC by vein weekly and Radiation Therapy 63 GY/35 fractions for 7 weeks cycles
  Interventions: Drug: Erlotinib; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Erlotinib — 150 mg by mouth daily for 7 Weeks
  Other Names: Tarceva; OSI-774; Erlotinib Hydrochloride
Drug: Carboplatin — 2 AUC by vein weekly for 7 Weeks
  Other Names: Paraplatin
Drug: Paclitaxel — 45 mg/m^2 by vein weekly for 7 Weeks
  Other Names: Taxol
Radiation: Radiation Therapy — 63 GY/35 fractions for 7 weeks (+/- 5 days)
  Other Names: RT; Radiotherapy

SUMMARY:
The goal of this clinical research study is to find out if erlotinib given with chemotherapy and radiation therapy can help to control NSCLC. The safety of this combination treatment will also be studied.

Researchers will also test the tissue from your earlier biopsy to measure the levels of epidermal growth factor receptor (EGFR). The purpose of EGFR testing is to learn about any link between various forms of EGFR and your response to treatment with erlotinib.

DETAILED DESCRIPTION:
Erlotinib is designed to block the activity of a protein called epidermal growth factor (EGFR). EGFR is found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a FEV1 (breathing test). You will have a complete physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate). Blood (about 2 tablespoons) will be drawn for routine tests. You will have a computed tomography (CT) scan or magnetic resonance imaging (MRI) of the brain to check the status of the disease. You will be required to have a positron emission tomography (PET) scan to locate the area of cancer outside the chest and lymph glands. You will have either a CT scan or an MRI to measure the size of the tumor(s). If there is positive finding of CT or MRI you will be taken off study. You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart). If you have a significant history of cardiovascular disease, you will have a MUGA scan and echocardiogram to test your heart function. Women who are able to have children must have a negative urine or blood (about 2 teaspoons) pregnancy test before starting treatment.

You will have PET scan 1 month after completion of consolidation chemotherapy.

If you are found to be eligible to take part in this study, you will take erlotinib every day for 7 weeks (except on the days you receive chemotherapy). The erlotinib tablets should be taken at the same time each day, at least 1 hour before or 2 hours after a meal, with a small glass (about 7 ounces) of water. If you are unable to swallow tablets, you may dissolve the tablets in distilled water to drink.

You will receive radiation every day (Monday through Friday) for 7 weeks. You will also receive chemotherapy through a needle in a vein once a week for 7 weeks. The chemotherapy will include carboplatin and paclitaxel. Receiving chemotherapy will take about 6 hours total.

You will receive consolidation therapy on weeks 11-17.

Treatment on this study will last 17 weeks. Once a week during that time, you will have blood (about 2 tablespoons) drawn for routine tests. You will also have a CT scan of the chest within about 4 weeks from beginning the study, 2 months after finishing therapy, and then every 6 months after that for 2 years. The CT scans are used to check the status of the disease.

You will be taken off study if the disease gets worse or intolerable side effects occur. In this case, you would not receive erlotinib anymore but would continue standard chemotherapy and radiation therapy.

You will be asked to come in to the clinic for follow-up visits to check on your recovery from treatment. The follow-up visits will be at the end of all treatment, 1 month after treatment, and then once a month for as long as your doctor feels it is necessary. Once your side effects have become less severe, you will be asked to come in to the clinic for follow-up visits every 3 months for 2 years, and then every 4 months for the following 2 years after that. You will have a physical exam, and your medical history will be recorded. You will be asked about any side effects you may have. Blood (about 2 tablespoons) will be drawn for routine tests. You will have a PET scan.

You have the right to leave the study at any time. If you choose to stop participating in this study, you should contact the study chair and/or research nurse. Your doctor may decide to take you off this study if your medical condition gets worse and/or you are unable to comply with study requirements.

At the end of the study you will not be automatically notified of the research findings. If you wish to learn about the results, however, you may request them from the study chair.

This is an investigational study. All three study drugs are commercially available. Carboplatin, and paclitaxel are FDA approved for the treatment of NSCLC, but their use in combination with erlotinib is not. Erlotinib is FDA approved for some uses, but it has not been approved by the FDA to treat lung cancer patients like yourself who have not yet undergone chemotherapy; however, the FDA has permitted its use in this research study. Carboplatin and paclitaxel are considered standard of care treatment and you would probably be treated with these drugs or similar drugs even if you decided not to be in the study. Up to 48 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented NSCLC, including squamous cell carcinoma, adenocarcinoma (including bronchoalveolar cell), and large cell anaplastic carcinoma (including giant and clear cell carcinomas) and poorly differentiated (not otherwise specified, NOS) non-small cell lung cancer; totally resected tumors are excluded. ·
2. Patients must be M0;
3. Patients with Tl or T2 disease with N2 or T3N1-2 disease (Stage IIIA) are eligible if they are deemed inoperable. Patients with T4 with any N or any T with N2 or N3 disease are eligible if unresectable. Radiographic evidence of mediastinal lymph nodes > 2.0 cm in the largest diameter is sufficient to stage N2 or N3 disease. If the largest mediastinal node is < 2.0 cm in diameter and this is the basis for stage III disease, then at least one of the nodes must be proven positive cytologically or histologically;
4. Measurable disease is required
5. Patients with tumors adjacent to a vertebral body are eligible as long as all gross disease can be encompassed in the radiation boost field. The boost volume must be limited to < 50% of the ipsilateral lung volume.
6. Patients must be greater than or equal to 18 years of age;
7. Patients with Zubrod performance status 0-1
8. Adequate hematologic function defined as: ANC greater than or equal 1,500/mm^3, platelets greater than or equal 100,000/mm^3, and hemoglobin greater than or equal 9 g/dL (prior to transfusions); adequate hepatic function defined as: total bilirubin less than or equal to 1.5 mg/dl, SGOT or SGPT less than or equal to 3 x ULN, adequate renal function defined as a serum creatinine level less than or equal to 2.0 mg/dl, alkaline phosphatase less than or equal to 2.5 x ULN, glucose less than or equal to 2 x ULN;
9. FEV1 with greater than or equal to 1000 cc;
10. Patients with weight loss less than or equal to than </= 10% over the past 3 months;
11. Patients with a pleural effusion that is a transudate, cytologically negative and nonbloody are eligible if the radiation oncologists feel the tumor can still be encompassed within a reasonable field of radiotherapy. If a pleural effusion can be seen on the chest CT but not on CXR and is too small to tap, the patient is eligible.
12. If patients had exploratory thoracotomy, they must have recovered from the procedure. Exploratory Thoracotomy and beginning of treatment should be within one month.
13. Women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]) and male participants must practice effective contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study and for four weeks after completion of treatment.
14. For women of childbearing potential, a urine or blood pregnancy test must be performed within 48 hours prior to the start of protocol treatment;
15. Medical Oncology and Radiation Oncology consults and approval.
16. Patients must sign a study-specific consent form prior to study entry.

Exclusion Criteria:

1. Prior systemic chemotherapy and/or thoracic radiotherapy for any reason and/or surgical resection of present cancer;
2. Exudative, bloody, or cytologically malignant effusion or effusion that are exudative and/or bloody and are suggestive or malignant involvement.
3. Prior therapy with any other drug that targets the EGFR pathway,
4. Active pulmonary infection not responsive to conventional antibiotics;
5. History of interstitial lung disease;
6. History of severe COPD requiring greater than or equal to 3 hospitalizations over the past year;
7. Significant history of cardiac disease, i.e., uncontrolled hypertension, unstable angina, uncompensated congestive heart failure, myocardial infarction within the past year, or cardiac ventricular arrhythmias requiring medication; patients with left ventricular ejection fraction (LVEF) below the institutional range of normal (50-70%) on a baseline multiple gated acquisition (MUGA) scan or echocardiogram.
8. Patients with > grade 1 neuropathy;
9. Evidence of malignancy in the past 3 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other in situ cancers;
10. Women who are pregnant or breast feeding, as treatment involves unforeseeable risks to the participant, embryo, fetus, or nursing infant; women with a positive pregnancy test on enrollment or prior to study drug administration;
11. Women of childbearing potential and male participants who are unwilling or unable to use an acceptable method of contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study and for four weeks after completion of treatment or those who are using a prohibited contraceptive method (methods with unknown efficacy).
12. Patients who currently are participating in other clinical trials and/or who have participated in other clinical trials in the previous 30 days. Clinical trials involving administration of investigational agents or interfering with the safe conduct of this trial. All clinical trials would exclude observational trials which would not interfere with the endpoints of our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Lin, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Komaki R, Allen PK, Wei X, Blumenschein GR, Tang X, Lee JJ, Welsh JW, Wistuba II, Liu DD, Hong WK. Adding Erlotinib to Chemoradiation Improves Overall Survival but Not Progression-Free Survival in Stage III Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2015 Jun 1;92(2):317-24. doi: 10.1016/j.ijrobp.2015.02.005. PMID 25968826
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period: Nov 20, 2007 to June 18,2010. Total 68 stage IIIA/IIIB Non-Small Cell Lung Cancer (NSCLC) patients registered in the study. Eligible criteria: stage III NSCLC, inoperable, Karnofsky score ≥ 80, weight loss ≤5% in 3 months, forced expiratory volume in 1 second ≥ 1.0 L, and adequate hematologic, hepatic, and renal function.
Pre-assignment Details: There were 20 patients off-study after enrollment due to screen failure. Two patients were taken off protocol: 1 for diarrhea unrelated to treatment and the other for chemotherapy-induced chest pain. Only 46 patients are evaluable for this study.
Groups:
- Phase II TARCEVA (Erlotinib) With Chemoradiation in Stage IIIA: TARCEVA (erlotinib) 150 mg, P.O., daily, except for chemotherapy. Paclitaxel, 45mg/m2; Carboplatin, AUC=2, weekly; RT: 63Gy/35 fractions/7 weeks
Period: Overall Study
Arm/Group | Phase II TARCEVA (Erlotinib) With Chemoradiation in Stage IIIA
Started | 68
Completed | 46
Not Completed | 22
Not completed — Withdrawal by Subject | 2
Not completed — Screen Failures | 20

BASELINE CHARACTERISTICS:
Population: 48 patients registered and treated under the protocol.
Arm/Group | Phase II TARCEVA (Erlotinib) With Chemoradiation in Stage IIIA
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 23
Age, Continuous [Median (Full Range); unit: years] | 63.5 [46 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 42
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 46
  Mexico | 1
  United Arab Emirates | 1
Participants characteristic for completed treatment under the protocol and evaluable [Number; unit: participants] — Disease stage by American Joint Committee on Cancer [AJCC] 6th Ed:
  Stage IIIA: T1-3 N2 M0, Stage IIIB: T1-2 N3 M0 (contralateral mediastinal LN) or T4 Nx M0 (primary tumor involving mediastinal structures).
  The earlier TNM staging, the better treatment outcome. The KPS:100 is "perfect" Normal health, 90 is able to carry on normal activity, minor signs or symptoms of disease, and 80 is normal activity with effort; some signs or symptoms of disease. The KPS was to allow physicians to evaluate a patient's survival. The higher KPS scores, the better treatment outcome.
  participants
    Disease Stage IIIA | 22
    Disease Stage IIIB | 26
    Tumor Histology Adenocarcinoma | 23
    Tumor Histology Squamous Cell Carcinoma | 15
    Tumor Histology NSCLC Unspecified | 9
    Karnofsky performance score (KPS) 100 | 3
    Karnofsky performance (KPS) score 90 | 32
    Karnofsky performance(KPS) score 80 | 13
    EGFR status Wild-type | 38
    EGFR status- Mutated or deleted | 4
    EGFR status Unknown | 6
    Smoking history Former | 36
    Smoking history Current | 6
    Smoking history Never | 6
    Tumor HistologyLarge Cell Neuroendocrine Carcinoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Time To First Disease Progression
Description: Primary Endpoints is efficacy of concurrent erlotinib and chemoradiation as measured by time to progression. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions. All patients will be evaluated by followed up one month after treatment, once a month until recovery from treatment related toxicities, then every 3 months for 2 years, then every 4 months for 2 years (total of 4 years), then annually up to 5 years.
Time Frame: From date of registration until the date of first documented progression or death from any cause, or lost to follow up, whichever came first, assessed up to 5 years.
Population: There were 46 out of 48 patients completed treatment under the protocol and evaluable for data analysis. 2 patients cannot complete the treatment and off-study. 1 for diarrhea unrelated to treatment and the other for chemotherapy-induced chest pain.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Phase II TARCEVA (Erlotinib) With Chemoradiation in Stage IIIA
Number analyzed (Participants) | 46
Month | 14 [9.0 to 18.6]

2. Secondary Outcome: Overall Survival and Disease Local Control Rate
Description: The Secondary Endpoints is Overall Survival (OS)and Disease Local Control (DLC)Rate. All patients will be followed up to evaluate Overall Survival and Disease Local Control by one month after treatment, once a month until recovery from treatment related toxicities, then every 3 months for 2 years, then every 4 months for 2 years (total of 4 years), then annually up to 5 years.
  CT scan of the chest/upper abdomen, MRI of brain or CT, and/or PET scan images are recommended to confirm the recurrence.
  Survival endpoints were estimated using the Kaplan-Meier method.
Time Frame: OS: From date of registration until the date of first documented death or lost to follow up, whichever came first, accessed up to 5 years. DLC: From date of registration until the date of first documented local disease recurrence, accessed up to 5 years.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Phase II TARCEVA (Erlotinib) With Chemoradiation in Stage IIIA
Number analyzed (Participants) | 46
percentage of participants
  Overall Survival:5-year | 35.9
  Disease Free Survival:5-year | 25.8
  Local Regional Survival:5-year | 55.8
  Distant Metastasis Free Survival:5-year | 36.5

ADVERSE EVENTS:
Time Frame: From the time of registration through study completion and follow up, assessed up to 5 years.
Arm/Group | Phase II TARCEVA (Erlotinib) With Chemoradiation in Stage IIIA
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 10/46
Other Adverse Events (participants affected / at risk) | 36/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II TARCEVA (Erlotinib) With Chemoradiation in Stage IIIA (N=46)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Pneumonititis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Skin toxicity, any (Skin and subcutaneous tissue disorders) | 6 (6)
Acneform rash (Skin and subcutaneous tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II TARCEVA (Erlotinib) With Chemoradiation in Stage IIIA (N=46)
Esophagitis (Gastrointestinal disorders) | 18 (18)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Skin toxicity, any (Skin and subcutaneous tissue disorders) | 10 (10)
Acneform rash (Skin and subcutaneous tissue disorders) | 28 (28)
Fatigue (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT00563784/Prot_SAP_000.pdf